CLINICAL TRIAL: NCT01933984
Title: Individualized Dosing Schedule of Inhaled Bronchodilator for Endotracheally Intubated Chronic Obstructive Pulmonary Disease Patients
Brief Title: Individualized Dosing Schedule of Inhaled Bronchodilator for Endotracheally Intubated COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin-hwar Wu (Other)
Responsible Party: Sponsor-Investigator, Shin-hwar Wu, Attending physician, Changhua Christian Hospital
Organization: Changhua Christian Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102-CCH-IRP-017
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Bronchodilator agents,; chronic obstructive pulmonary disease,; endotracheal intubation,; mechanical ventilator
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate; Fluticasone; Fenoterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized dosing (Experimental): * Ventilator support
  * Determining personal target airway resistance
  * Bronchodilator:Salmeterol/fluticasone 4 puffs inhalation every 12 hours until ventilator discontinuation or the 28th day if ventilator-dependent
  * Bronchodilator:Ipatropium/salbutamol 1 vial inhalation every 6 hours for the first 3 days
  * Steroid:Methylprednisolone 40 mg intravenous injection every 8 hours for the first 3 days
  * Additional broncho-dilators inhalation: Salmeterol/fluticasone (Seretide) 4 puffs plus fenoterol (Berotec) 4 puffs inhalation if personal target airway resistance (measured every 8 hours) not met (until ventilator discontinuation or the 28th day if ventilator-dependent)
  Interventions: Drug: Bronchodilators inhalation
- Fixed dosing (Active Comparator): * Ventilator support
  * Determining personal target airway resistance
  * Bronchodilator:Salmeterol/fluticasone 4 puffs inhalation every 12 hours until ventilator discontinuation or the 28th day if ventilator-dependent
  * Bronchodilator:Ipatropium/salbutamol 1 vial inhalation every 6 hours for the first 3 days
  * Steroid:Methylprednisolone 40 mg intravenous injection every 8 hours for the first 3 days
  * No additional bronchodilator given if personal target airway resistance (measured every 8 hours) not met
  Interventions: Drug: Bronchodilators inhalation

INTERVENTIONS:
Drug: Bronchodilators inhalation — Salmeterol/fluticasone (Seretide Evohaler) 4 puffs plus fenoterol (Berotec)(0.1mg/puff) 4 puffs inhalation when target airway resistance, measured every 8 hours, not met
  Other Names: Salmeterol/fluticasone (Seretide Evohaler); fenoterol (Berotec)(0.1mg/puff)

SUMMARY:
This study evaluates whether individualized dosing schedule of inhaled bronchodilator is more effective than fixed dosing in reducing airway resistance of intubated COPD patients.

DETAILED DESCRIPTION:
*Study Design

* This is an open-label, randomized controlled study comparing individualized versus fixed bronchodilator dosing schedule for patients with COPD with acute respiratory failure.

  *Patients Enrollment
* We will collect 100 patients just admitted to the intensive care unit of Changhua Christian Hospital (Changhua, Taiwan) due to COPD with acute respiratory failure.All participants will be randomly assigned to either group according to a computer-generated allocation sequence in block size of 4 patients.

  *Airway Resistance (Raw) Determination
* Enrolled patients will be ventilated by either AVEA (CareFusion, Yorba Linda, CA, USA),e500 (Newport Medical Instrument Inc. CA, USA) or Eivta 4 (Drager) ventilator. When evaluating Raw, the ventilator settings will be transiently switched to volume control mode with fixed tidal volume (500 ml) and constant flow (with a rate of 60 L/min). Plateau pressure is measured by manually controlled end-inspiratory pause12. Every effort will be exercised to avoid excessive airway secretion or patient agitation during measurement. Each measurement will be repeated three times with an interval of at lease 1 minute and calculate their average. Raw will be calculated by an equation of (peak inspiratory pressure - plateau pressure)/flow. After each measurement, the ventilator will soon be reverted to its usual settings. Raw will be routinely determined every 8 hours for 28 days if the ventilator is not discontinued.

  *Technique of Metered Dose Inhaler (MDI) administration through endotracheal tube
* The technique basically follows the recommendation of Dhand and Guntur. Airway secretions should be sucked out before drug administration. Heat moisture exchanger, but not humidifier, is removed. After shaking and warming MDI to hand temperature, the canister is connected to an AeroChamber HC MV spacer (Trudell Medical International, London, Canada) placed in the inspiratory limb of ventilator circuit 15 cm away from the endotracheal tube. Actuation is synchronized with the initiation of inspiration. Each actuation is at least 15 second apart.

  *Personal Target Raw Determination
* The target Raw of each patient should be determined within 72 hours after their admission to intensive care unit. After confirming no inhaled bronchodilator given in preceding 2 hours (for fenoterol) or 12 hours (for salmeterol/fluticasone), we will deliver 3 consecutive doses of 4 puffs, 8 puffs and 16 puffs of fenoterol MDI (100 mcg/puff, Berotec;Boehringer Ingelheim, Ingelheim, Germany) inhalation with each dose 15 minutes apart. The Raw measured 15 minutes later is assigned as this patient's personal target Raw.

  *Bronchodilator Delivery Schedule
* Each patient will routinely receive 4 puffs of 25 mcg salmeterol /250 mcg fluticasone (Seretide Evohaler 250; GlaxoSmithKline Inc. Evreux, France) every 12 hours until the discontinuation of ventilator. Each patient will also routinely receive 1 vial of Combivent (ipatropium bromide 0.5 mg and salbutamol sulfate 2.5 mg) every 6 hours and be injected with intravenous methylprednisolone 40mg every 8 hours in the initial 3 days.The use of short acting bronchodilator in an as-needed basis is not restricted. According to the Raw data determined every 8 hours, individualized dosing group will receive an additional 4 puffs of 25 mcg salmeterol /250 mcg fluticasone plus 4 puffs of fenoterol if the value is higher than personal target Raw (Once it coincides with regular dosing period of salmeterol/fluticasone, only fenoterol will be added). No such extra dose will be given to fixed dosing (control) group regardless of Raw value.

  *Statistical Analysis
* Student's t test will be used to compare ∆Raw of both groups. For the comparisons of other continuous variables without distribution normality, Wilcoxon rank sum test will be used. When comparing two categorical variables, Chi-square or Fisher's exact test will be used when appropriate. A P value of less than 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* chronic obstructive pulmonary disease
* acute respiratory failure under ventilator support for less than 72 hours
* endotracheal tube inserted

Exclusion Criteria:

* confirmed asthma
* Acute Physiology and Chronic Health Evaluation II score over 35
* a co-morbidity of septic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-08; Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shin-hwar Wu, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan, China

IPD SHARING:
Plan to Share IPD: No
We have no plan to share IPD.

REFERENCES:
- [Background] Fuller HD, Dolovich MB, Posmituck G, Pack WW, Newhouse MT. Pressurized aerosol versus jet aerosol delivery to mechanically ventilated patients. Comparison of dose to the lungs. Am Rev Respir Dis. 1990 Feb;141(2):440-4. doi: 10.1164/ajrccm/141.2.440. PMID 2154154
- [Background] Aerosol consensus statement. Consensus Conference on Aerosol Delivery. Chest. 1991 Oct;100(4):1106-9. No abstract available. PMID 1914568
- [Background] Dhand R, Duarte AG, Jubran A, Jenne JW, Fink JB, Fahey PJ, Tobin MJ. Dose-response to bronchodilator delivered by metered-dose inhaler in ventilator-supported patients. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):388-93. doi: 10.1164/ajrccm.154.2.8756811.
- [Background] Naranjo CA, Busto U, Sellers EM, Sandor P, Ruiz I, Roberts EA, Janecek E, Domecq C, Greenblatt DJ. A method for estimating the probability of adverse drug reactions. Clin Pharmacol Ther. 1981 Aug;30(2):239-45. doi: 10.1038/clpt.1981.154. No abstract available. PMID 7249508
- [Background] Malliotakis P, Linardakis M, Gavriilidis G, Georgopoulos D. Duration of salmeterol-induced bronchodilation in mechanically ventilated chronic obstructive pulmonary disease patients: a prospective clinical study. Crit Care. 2008;12(6):R140. doi: 10.1186/cc7117. Epub 2008 Nov 14. PMID 19014570
- [Derived] Wu SH, Shyu LJ, Li CH, Yu CH, Chen HC, Kor CT, Wang CH, Lin KH. Better airway resistance reduction profile in intubated COPD patients by personalized bronchodilator dosing: A pilot randomized control trial. Pulm Pharmacol Ther. 2018 Apr;49:134-139. doi: 10.1016/j.pupt.2018.02.004. Epub 2018 Feb 21. PMID 29474893

RESULTS

PARTICIPANT FLOW:
Groups:
- Individualized Dosing: * Ventilator support
  * Determining personal target airway resistance
  * Salmeterol/fluticasone 4 puffs inhalation q12h until ventilator discontinuation or the 28th day if ventilator-dependent
  * Ipatropium/salbutamol 1 vial inhalation q6h for the first 3 days
  * Methylprednisolone 40 mg intravenous injection q8h for the first 3 days
  * Additional Salmeterol/fluticasone (Seretide) 4 puffs plus fenoterol (Berotec) 4 puffs inhalation if personal target airway resistance (measured every 8 hours) not met
- Fixed Dosing: Ventilator support
  * Determining personal target airway resistance
  * Salmeterol/fluticasone 4 puffs inhalation q12h until ventilator discontinuation or the 28th day if ventilator-dependent
  * Ipatropium/salbutamol 1 vial inhalation q6h for the first 3 days
  * Methylprednisolone 40 mg intravenous injection q8h for the first 3 days
  * No additional bronchodilator given if personal target airway resistance (measured every 8 hours) not met
Period: Overall Study
Arm/Group | Individualized Dosing | Fixed Dosing
Started | 26 | 25
Completed | 26 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individualized Dosing | Fixed Dosing | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (13.3) | 77.9 (8.7) | 75.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 21 | 23 | 44
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 26 | 25 | 51
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.6 (11.6) | 23.4 (4.9) | 24.5 (8.9)

OUTCOME MEASURES:

1. Primary Outcome: ∆Raw (the Difference Between Measured and Target Airway Resistance)
Description: The value can be expressed as relative deviation from target =(measured Raw - target Raw)/target Raw X100
Time Frame: Airway resistance will be recorded everyday. If a patient's ventilator was liberated less than 28 days, the day of liberation was the reported time frame. If the day of ventilator liberation was over 28 days, the 28th day was the reported time frame.
Population: The deviation of Raw from the personal target, which was calculated as (measured Raw-target Raw)/target Raw.
Measure: Mean (Standard Deviation); unit: percentage of relative Raw deviation
Groups:
- Individualized Dosing: * Ventilator support
  * Determining personal target airway resistance
  * Bronchodilator:Salmeterol/fluticasone 4 puffs inhalation every 12 hours until ventilator discontinuation or the 28th day if ventilator-dependent
  * Bronchodilator:Ipatropium/salbutamol 1 vial inhalation every 6 hours for the first 3 days
  * Steroid:Methylprednisolone 40 mg intravenous injection every 8 hours for the first 3 days
  * Additional broncho-dilators inhalation: Salmeterol/fluticasone (Seretide) 4 puffs plus fenoterol (Berotec) 4 puffs inhalation if personal target airway resistance (measured every 8 hours) not met (until ventilator discontinuation or the 28th day if ventilator-dependent) salmeterol/fluticasone: Each puff contains 25 mcg salmeterol /250 mcg fluticasone ipatropium/salbutamol: Each vial contains ipatropium bromide 0.5 mg and salbutamol sulfate 2.5 mg Methylprednisolone Additional broncho-dilators inhalation: Salmeterol/fluticasone (Seretide Evohaler) 4 puffs plus fenoterol (Berotec)(0
- Fixed Dosing: * Ventilator support
  * Determining personal target airway resistance
  * Bronchodilator:Salmeterol/fluticasone 4 puffs inhalation every 12 hours until ventilator discontinuation or the 28th day if ventilator-dependent
  * Bronchodilator:Ipatropium/salbutamol 1 vial inhalation every 6 hours for the first 3 days
  * Steroid:Methylprednisolone 40 mg intravenous injection every 8 hours for the first 3 days
  * No additional bronchodilator given if personal target airway resistance (measured every 8 hours) not met salmeterol/fluticasone: Each puff contains 25 mcg salmeterol /250 mcg fluticasone ipatropium/salbutamol: Each vial contains ipatropium bromide 0.5 mg and salbutamol sulfate 2.5 mg Methylprednisolone Determining personal target airway resistance: Three consecutive doses of 4, 8 and 16 puffs of fenoterol MDI (100 mcg/puff, Berotec;Boehringer Ingelheim, Ingelheim, Germany) inhalation with each dose 15 minutes apart. The airway resistance measured 15 minutes later is assigned as th
Arm/Group | Individualized Dosing | Fixed Dosing
Number analyzed (Participants) | 26 | 25
percentage of relative Raw deviation | 9 (10) | 44 (11)

2. Primary Outcome: Rapidity of ∆Raw Change
Description: The deviation of ∆Raw from the personal target, which was calculated as (measured Raw-target Raw)/target Raw multiplied by 100.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of relative Raw deviation
Arm/Group | Individualized Dosing | Fixed Dosing
Number analyzed (Participants) | 26 | 25
percentage of relative Raw deviation | -3 (9.7) | 0.4 (13.9)

3. Secondary Outcome: Ventilator-free Days From Day 1 to 28
Description: Ventilator-free days from day 1 to 28 after enrollment
Time Frame: From day 1 to day 28 after enrollment
Measure: Number; unit: day
Arm/Group | Individualized Dosing | Fixed Dosing
Number analyzed (Participants) | 26 | 25
day | 19 | 22

4. Secondary Outcome: The Participants of Breathing Without Assistance by Day 28
Description: The number of participants who breath without ventilator by day 28
Time Frame: the 28th day after enrollment
Measure: Number; unit: the number of participants
Arm/Group | Individualized Dosing | Fixed Dosing
Number analyzed (Participants) | 26 | 25
the number of participants | 19 | 22

5. Secondary Outcome: Number of Episode of Nosocomial Pneumonia
Description: The number of episodes of nosocomial pneumonia happened by day 28. And nosocomial pneumonia is a lower respiratory infection that was not incubating at the time of hospital admission and that presents clinically 2 or more days after hospitalization.
Time Frame: the 28th day after enrollment
Measure: Median (Standard Deviation); unit: episodes of nosocomial pneumonia
Arm/Group | Individualized Dosing | Fixed Dosing
Number analyzed (Participants) | 26 | 25
episodes of nosocomial pneumonia | 0 (0) | 0 (0)

6. Secondary Outcome: Number of Total Puff of Rescue Short-acting Bronchodilator
Description: The number of total puff of rescue short-acting bronchodilator.
Time Frame: the 28th day after enrollment
Measure: Number; unit: puffs
Arm/Group | Individualized Dosing | Fixed Dosing
Number analyzed (Participants) | 26 | 25
puffs | 0 | 0

7. Secondary Outcome: Numbers of Episode of Drug-related Adverse Effect
Description: The numbers of episode of drug-related adverse effect. Naranjo score should be over 4 to be considered drug-related adverse effect. Naranjo score range form 0 to 9, and the higher scores means a higher relationship with drug-related adverse effect.
Time Frame: From day 1 to day 28 after enrollment
Measure: Median (Standard Deviation); unit: episodes
Arm/Group | Individualized Dosing | Fixed Dosing
Number analyzed (Participants) | 26 | 25
episodes | 0 (0) | 0 (0)

8. Secondary Outcome: Mortality Rate
Description: The percentage of participants died at day 180.
Time Frame: the 180th day after enrollment
Measure: Number; unit: percentage of participants
Arm/Group | Individualized Dosing | Fixed Dosing
Number analyzed (Participants) | 26 | 25
percentage of participants | 35 | 40

ADVERSE EVENTS:
Time Frame: From day 1 to day 28
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, are same with the clinicaltrials.gov definitions. However, only events with Naranjo score over 4 were be considered as drug-related.
  No treatment-related adverse events could be found in this study. So, no additional information could be offered.
Arm/Group | Individualized Dosing | Fixed Dosing
All-Cause Mortality (participants affected / at risk) | 9/26 | 10/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-05-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT01933984/Prot_SAP_000.pdf